CLINICAL TRIAL: NCT02305875
Title: The Musculocutaneous Nerve (Mcn) in a High Resolution MRI
Brief Title: The Musculocutaneous Nerve in a High Resolution MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Trygve Kjelstrup, MD, Section manager, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-04115B
Record Dates: First submitted 2014-11-19; First posted 2014-12-03 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Brachial Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCN scoring (Experimental): Scoring of the mcn nerve's position in the axillary sheat using MRI
  Interventions: Other: MCN scoring

INTERVENTIONS:
Other: MCN scoring — Mcn's distance from top of the humeral head. Mcn's distance to the catheters insertion point. Mcn's distance and position in relationship to the axillary artery.

SUMMARY:
The investigators have made a favourable experience with the in 2006 published transarterial triple injection method [4]. This classic method combines the block effect of an axillary catheter injection (median nerve position) with a double transarterial injection at terminal nerve level in the axilla.

The investigators experience after a recent published MRI study [3], confirms that a proximal axillary local anesthetic injection via an axillary catheter, guided by nerve stimulator, is beneficial for the block effect. The MRI study was conducted using nerve stimulation and a transarterial technique. The proximal injection with an effect at cord level, combined with axillary injections at terminal nerve level, produce an effective block distal to the elbow.

The proximal injection has obviously an effect to the lateral cord and the musculocutaneous nerve (mcn) [3]. Recent studies have advocated that a double axillary injection method is sufficient for the axillary block [5, 6]. Their block techniques included a selective block of the mcn at terminal nerve level. The investigators MRI study [3] demonstrated a successful block effect (analgesia or anaesthesia) of the mcn nerve in all patients (15 of 15 patients) in the triple injection group without a selective block of this nerve. In the 1- deposit (catheter injection) and 2-deposit (transarterial injections) group, 11 of 15 patients (73%) had the mcn successful blocked.

The objective in this study (Article 4) is to examine the mean position of the mcn nerve and its relationship to the coracobrachial muscle. Can MRI indicate / predict that a proximal directed axillary catheter in median nerve position is beneficial in order to provide a successful mcn blockade? Is a selective injection to the mcn at terminal nerve level superfluous when a catheter is used?

DETAILED DESCRIPTION:
45 patients were examined with MRI in a previous study [3] and now they underwent an additionally examination with a special focus on the anatomy and course of the mcn nerve. A line was drawn from the most cranial part of the humeral head perpendicular towards the brachial plexus. The distance from this line to the point where the mcn nerve entered the coracobrachial muscle was measured. This entering point was defined as the point where the mcn nerve left the axillary sheat. The visulaity of the mcn was scored as 0 = not visible, 1 = partly visible and 2 = clear visible.

The evaluation was a consensus assessment where all authors evaluated the T2-weighted, fat suppressed MRI images at the same time. If the mcn nerve could not be identified, the patients were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hand surgery
* ASA 1 - 2
* Weight from 50 - 95 kg
* MR compatible, suitable

Exclusion Criteria:

* Neurologic deficit
* Reaction to LA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Position of the musculocutaneous nerve in the axillary sheat. Mean distance in cm to the humeral head and the insertion point of the catheter in 54 patients. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Kr Hol, PhD, Study Director — University of Oslo, The Intervention Centre
Locations (1):
- The Intervention Centre, Rikshospitalet, Oslo University Hospital, Oslo, Norway